CLINICAL TRIAL: NCT04808401
Title: Influence of Different Inspired Oxygen Fractions on Perioperative Myocardial Biomarkers, Myocardial Strain and Outcome in Patients Undergoing General Anaesthesia for Elective Non-cardiac Surgery: A Prospective Randomized Open-label Single Centre Pilot Study
Brief Title: Influence of Oxygen on Perioperative Outcome in Patients Undergoing General Anaesthesia for Elective Non-cardiac Surgery
Acronym: Promise-O2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2020_02560
Record Dates: First submitted 2021-03-15; First posted 2021-03-22 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Coronary Artery Disease; Anesthesia
Keywords: Coronary Artery Disease; Transesophageal Echocardiography (TEE); Hyperoxia; Strain; Myocardial biomarkers; Normoxaemia; Anaesthesia
MeSH Terms: conditions — Coronary Artery Disease; Hyperoxia; Sprains and Strains | interventions — Oxygen

STUDY DESIGN:
Intervention Model Description: Patients start with a crossover design undergoing both TEE images at normoxia and hyperoxia in random order and then are randomized a second time to receive either normoxia or hyperoxia for the remaining procedure in a parallel design.
Who Masked: Outcomes Assessor
Masking Description: TEE images will be coded and analysed in batches at a later date by a blinded reader
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Normoxaemia First + Hyperoxia Procedure (Experimental): Patients will undergo TEE imaging at normoxaemia (FiO2=0.3) first, and hyperoxia (FiO2=0.8) will be targeted second. After the image acquisition patients receive hyperoxic concentrations.
  Interventions: Drug: Oxygen
- Normoxaemia First + Normoxia Procedure (Experimental): Patients will undergo TEE imaging at normoxaemia (FiO2=0.3) first, and hyperoxia (FiO2=0.8) will be targeted second. After the image acquisition patients receive normoxic concentrations.
  Interventions: Drug: Oxygen
- Hyperoxia First + Hyperoxia Procedure (Experimental): Patients will undergo TEE imaging at hyperoxia (FiO2=0.8) first, and normoxaemia (FiO2=0.3) will be targeted second. After the image acquisition patients receive hyperoxic concentrations.
  Interventions: Drug: Oxygen
- Hyperoxia First + Normoxaemia Procedure (Experimental): Patients will undergo TEE imaging at hyperoxia (FiO2=0.8) first, and normoxaemia (FiO2=0.3) will be targeted second. After the image acquisition patients receive normoxic concentrations.
  Interventions: Drug: Oxygen

INTERVENTIONS:
Drug: Oxygen — Two FIO2 settings during stable general anaesthesia resulting in normoxaemic and hyperoxic arterial oxygen partial pressures.
  Other Names: Medical gas

SUMMARY:
The purpose of this study is to investigate the impact of supraphysiologic oxygen (hyperoxia) on myocardial function in anaesthetized patients undergoing non-cardiac vascular surgery.

DETAILED DESCRIPTION:
Up to 110 patients with either proven coronary artery disease (CAD) or two or more risk factors for CAD undergoing elective or non-emergent non-cardiac vascular surgery will be recruited. Three blood samples for levels of myocardial biomarkers will be obtained at different perioperative time points (before anaesthesia induction, 2 hours after skin closure and 24 hours after the end of the surgery). The three myocardial biomarkers investigated are high-sensitive Troponin T (hsTnT), N-terminal (NT)-pro hormone BNP (NT-proBNP) and heart-type fatty acid binding protein (H-FABP). In the timeframe shortly after the induction of anaesthesia and prior to the start of surgery, myocardial strain as a marker of cardiac function will be measured by transesophageal echocardiography (TEE). Echocardiography measurements will be acquired at two different oxygen states for each patient.The fraction of inspired oxygen (FiO2) will be adjusted to reach a normoxaemic state (FiO2=0.3) and a hyperoxic state (FiO2=0.8). Patients will be randomized to which oxygen level is investigated first. Thereafter, the patients are again randomly assigned to either the normoxaemic or the hyperoxic state for the remainder of the perioperative treatment until 2 hours after skin closure. Surgery will be performed as planned by the treating team. Differences in the perioperative levels of myocardial biomarkers at the different time points and their dynamics will be assessed. Echocardiography images will be analyzed in a blinded manner for cardiac function and systolic and diastolic strain parameters. The results will help anaesthesiologists to better weigh risks and benefits when selecting an inspired oxygen fraction in such patients, and will help to evaluate hyperoxia as a risk factor for myocardial injury.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Patients eligible for the study should be scheduled for elective or non-emergent non-cardiac vascular surgery under general anaesthesia with endotracheal intubation, and have either
* proven CAD and will undergo high- or intermediate surgical risk procedure according to European (European Society of Cardiology, ESC / European Society of Anaesthesiology and Intensive Care, ESAIC) guidelines on non-cardiac surgery.

or

* two or more risk factors for CAD and will undergo high- or intermediate surgical risk procedures according to European ESC/ESAIC guidelines on non-cardiac surgery.

Exclusion Criteria:

* Acute coronary event 30 days before surgery
* Acute congestive heart failure
* Hemodynamic instability before induction of aneasthesia (vasopressor or inotrope infusion since hospitalization for index surgery)
* Atrial fibrillation or other severe arrhythmia
* Severe pulmonary disease (dependent on oxygen therapy or the Global Initiative for Chronic Obstructive Lung Disease (GOLD) stage 4 or severe carbon monoxide diffusion impairment or severe pulmonary hypertension)
* Preoperative oxygen saturation (SpO2) below 90% on room air
* Increased risk of oxygen toxicity (e.g., chemotherapy for malignancy within 3 months, bleomycin treatment, airway laser surgery)
* Scheduled surgery in the thoracic cavity
* ICU admission for respirator weaning and delayed extubation
* Pre-existing surgical site infection (SSI)
* Current active signs of systemic inflammatory response syndrome (SIRS) or sepsis according The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3)
* Pregnancy
* Emergency surgery (to be performed within less than 12 hours of scheduling)
* Ambulatory surgery
* Baseline hs-TnT level elevated above 65ng/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2021-05-07 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Difference in hsTnT from preoperative baseline | at 24 hours after surgery
  ng/L

SECONDARY OUTCOMES:
Incidence of myocardial injury in non-cardiac surgery (MINS) | at 24 hours after surgery
  MINS is defined as an absolute change of hsTnT levels of at least 5ng/L from preoperative baseline or an hs-TnT level of at least 65ng/L
Difference in high sensitive TnT from preoperative baseline | at 2 hours after surgery
  ng/L
Differences in N-terminal pro B-type natriuretic peptide (NT-proBNP) from preoperative baseline | at 2 hours and 24 hours after surgery
  pg/ml
Differences in heart type fatty acid binding protein (H-FABP) from preoperative baseline | at 2 hours and 24 hours after surgery
  pg/ml
Difference in myocardial time to peak strain between oxygen levels | Through study completion, within 1hour post-induction
  Milliseconds (ms)
Difference in myocardial strain rate between oxygen levels | Through study completion, within 1hour post-induction
  Change in strain over time (/second)
Difference in myocardial strain rate ratio between oxygen levels | Through study completion, within 1hour post-induction
  Change in E/A ratio
Difference in myocardial displacement between oxygen levels | Through study completion, within 1hour post-induction
  Millimeters (mm)
Difference in myocardial time to peak displacement between oxygen levels | Through study completion, within 1hour post-induction
  Milliseconds (ms)
Difference in myocardial velocities between oxygen levels | Through study completion, within 1hour post-induction
  Change in displacement over time (millimeters/second)
Difference in myocardial velocity ratio between oxygen levels | Through study completion, within 1hour post-induction
  Change in E/A ratio
Difference in peak twist | Through study completion, within 1hour post-induction
  Degrees (°)
Difference in peak torsion | Through study completion, within 1hour post-induction
  Degrees/centimeter (°/cm)
Difference in ejection fraction (EF) | Through study completion, within 1hour post-induction
  Percent (%)
Difference in chamber volumes | Through study completion, within 1hour post-induction
  Millilitres (ml)

CONTACTS AND LOCATIONS:
Overall Officials: Dominik P Guensch, MD, Principal Investigator — Bern University Hospital, Inselspital; Jan-Oliver Friess, MD, Principal Investigator — Bern University Hospital, Inselspital
Locations (1):
- Bern University Hospital, Inselspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guensch DP, Fischer K, Yamaji K, Luescher S, Ueki Y, Jung B, Erdoes G, Grani C, von Tengg-Kobligk H, Raber L, Eberle B. Effect of Hyperoxia on Myocardial Oxygenation and Function in Patients With Stable Multivessel Coronary Artery Disease. J Am Heart Assoc. 2020 Mar 3;9(5):e014739. doi: 10.1161/JAHA.119.014739. Epub 2020 Feb 22. PMID 32089047
- [Background] Devereaux PJ, Szczeklik W. Myocardial injury after non-cardiac surgery: diagnosis and management. Eur Heart J. 2020 May 1;41(32):3083-3091. doi: 10.1093/eurheartj/ehz301. PMID 31095334
- [Background] Friess JO, Mikasi J, Baumann R, Ranjan R, Fischer K, Levis A, Terbeck S, Hirschi T, Gerber D, Erdoes G, Schoenhoff FS, Carrel TP, Madhkour R, Eberle B, Guensch DP. Hyperoxia-induced deterioration of diastolic function in anaesthetised patients with coronary artery disease - Randomised crossover trial. BJA Open. 2023 Apr 27;6:100135. doi: 10.1016/j.bjao.2023.100135. eCollection 2023 Jun. PMID 37588173